CLINICAL TRIAL: NCT03176732
Title: Mechanisms for Individual Differences in Hypertension in Obstructive Sleep
Acronym: PISA-BP
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 823172; P01HL094307-06A1 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Sleep Apnea, Obstructive; Hypertension
Keywords: Sleep Apnea; Hypertension; Positive Airway Pressure; Blood Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — As a part of the research protocol, we intend to draw from each participant at baseline and following 4 months of PAP therapy. All samples will be processed according to the recommended procedures for the different analyses we intend to measure and stored at -80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Normotensive: Categorized by 24-hr systolic BP (SBP): normotensive (< 125 mm Hg) on no BP medications
  Interventions: Device: Positive Airway Pressure
- Group 2: Controlled Hypertensive: Categorized by 24-hr systolic BP (SBP): controlled hypertensive (< 130 mm Hg) on BP medication(s) and/or lifestyle modification
  Interventions: Device: Positive Airway Pressure
- Group 3: Uncontrolled Hypertensive: Categorized by 24-hr systolic BP (SBP): uncontrolled hypertensive (≥ 130 mm Hg) on 0-2 BP medications
  Interventions: Device: Positive Airway Pressure
- Group 4: Hypertensive: Categorized by 24-hr systolic BP (SBP): hypertensive (≥ 135 mm Hg) resistant to 3 or more BP medications ideally including a diuretic (resistant hypertension)
  Interventions: Device: Positive Airway Pressure

INTERVENTIONS:
Device: Positive Airway Pressure — Participants will use Positive Airway Pressure (PAP) treatment

SUMMARY:
Hypertension is a common consequence of obstructive sleep apnea (OSA). However, not all individuals with OSA have hypertension and there are major individual differences in blood pressure response to positive airway pressure treatment of OSA. This project is focused on determining the basis of these individual differences in blood pressure response to OSA and will evaluate the possible underlying reasons for these differences. The results will help clinicians to know whether or not to expect a reduction in blood pressure (BP) to OSA treatment in a given patient and thereby personalize patient management.

DETAILED DESCRIPTION:
We seek to assess the clinical determinants and molecular/genetic mechanisms underlying known individual differences in BP response to obstructive sleep apnea (OSA). This will result in a more personalized approach to BP management of OSA patients. Hypertension is a common consequence of OSA. Animal studies with cyclical intermittent hypoxia indicate that oxidative stress is likely the major mechanism, but cardiovascular response to arousals may also play a role. However, not all individuals with OSA have hypertension. Moreover, recent meta-analyses of treatment trials of OSA show major individual differences in BP response. The largest drop in BP with positive airway pressure (PAP) therapy for OSA is in patients with resistant hypertension taking three or more BP medications. This project is focused on determining the basis of these individual differences in BP response to OSA and PAP treatment. For Aim 1, we will assemble four groups of OSA subjects with: 1) no hypertension; 2) controlled hypertension on medications and/or lifestyle modifications; 3) uncontrolled hyper-tension despite one or two anti-hypertensive medications; and 4) resistant hypertension. We will assess reductions in BP with PAP therapy with mean nocturnal (sleep) arterial BP being the primary end-point. The prediction is that group 4 will show the largest fall in BP, even after controlling for relevant covariates, group 3 the next biggest fall, while groups 1 and 2 will show minimal BP changes. Both intent to treat and per protocol analyses, i.e., analyzing only those subjects who had PAP adherence of ≥ 4 hours/day and are adherent to medication, will be conducted. All subjects will have the following measured before and after 4 months of therapy: urinary isoprostanes and plasma levels of norepinephrine, renin activity, aldosterone, oxidized LDL, endothelin-1, and inflammatory biomarkers. In Aim 2, we hypothesize that those individuals with higher BP at baseline and the greatest BP response to PAP therapy will have higher levels of urinary isoprostanes and plasma norepinephrine at baseline and greater falls with therapy. Animal studies show that the key enzyme mediating oxidative stress in OSA is nicotinamide adenine dinucleotide phosphate-oxidase (NADPH) oxidase (NOX), in particular NOX2. Thus, NADPH oxidase activity will also be assessed. Individuals with the largest falls in BP on PAP therapy are hypothesized to have the highest activity of this enzyme at baseline. There are known genetic variants of this enzyme that affect its structure/activity. Thus, individual differences could be the result of genetic variants. To address this, we will employ in-depth sequencing and evaluate variants in 7 key genes regulating NOX2 structure/activity. Gene variants identified will be related to BP responses and to NADPH oxidase activity. In Aim 3, the role of arousals in the BP response to OSA will be assessed using a novel measurement of heart rate response to arousal. We hypothesize that the heart rate response to arousal will be related to the BP and molecular outcomes of Aims 1 and 2. Finally, given the complex relationship between OSA and BP, Aim 4 will utilize structural equation modeling to assess the relative impact of the various biological pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Apnea-Hypopnea Index (AHI) ≥ 15 events/hr on diagnostic polysomnography(PSG)
* No previous history of surgical treatment of OSA, and no medical treatment of OSA within the past 6 months
* Adherence to prescribed anti-hypertensive medications as assessed by an average adherence between Visits 1-2 of at least 0.85
* Arm circumference less than 50 cm

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* No telephone access or inability to return for follow-up
* Diagnosis of another sleep disorder in addition to OSA (e.g., periodic limb movement disorder [greater than 5 limb movements associated with arousal/hr of sleep], central sleep apnea [greater than 50% of apneas are central apneas], obesity hypoventilation syndrome, narcolepsy)
* Positive urine drug screen for any of the following: amphetamines, cocaine, opiates, barbiturates, benzodiazepines, phencyclidine (PCP), alcohol (ETOH), methadone (Visit 1)
* Requiring oxygen, bi-level positive airway pressure, or adaptive servo-ventilation for treatment of OSA
* Oxygen saturation < 87% for a period of 2 minutes during resting wakefulness during home sleep testing (HST) or PSG (Visit 2)
* Severe and inadequately controlled arterial hypertension (SBP greater than 180 mm Hg; diastolic BP greater than 110 mm Hg on 2 of 3 spot measurements on Visit 1)
* Participants with 24-hr SBP ≥ 140 mm Hg who are not on BP medications and participants on 4 or more BP medications with a 24-hr SBP < 135 mm Hg (Visit 2)
* A clinically unstable medical condition as defined by a change in medications in the previous month, including anti-hypertensive medications, or a new medical diagnosis in the previous 2 months (e.g., myocardial infarction, chronic heart failure, unstable angina, active infection, thyroid disease, depression or psychosis, cirrhosis, surgery, or cancer)
* Shift workers, individuals who regularly experience jet lag, or have irregular work schedules by history over the last 3 months
* Women who are pregnant or sexually active and of child-bearing age not using a form of contraceptive
* Routine consumption of > 2 alcoholic beverages/day Excessive use of caffeine (greater than 10 cups/day)
* Inability to communicate verbally or less than a 5th grade reading level

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects between the ages of 18 and 75 years of age with a diagnosis of untreated moderate to severe OSA as evidenced by an apnea/hypopnea index ≥ 15 events/hour who are about to be initiated on PAP treatment. We will make a conscious effort to recruit from all ethnic and social economic backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Nocturnal mean arterial blood pressure (nMAP) | Measured for 24-hours at baseline and repeated after 4 months of PAP treatment.
  Measured using 24-hour ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Oxidative stress | Collected overnight at baseline and repeated after 4 months of PAP treatment.
  Measured in urinary 8-isoprostane.
Sympathetic activity | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma

OTHER OUTCOMES:
Plasma renin | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma
Aldosterone | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma
Oxidized LDL | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma
Plasma endothelin-1 | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma
Inflammatory biomarkers | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood plasma
Neutrophil NADPH oxidase activity | Fasting blood draw collected at baseline and repeated after 4 months of PAP treatment.
  Measured in blood neutrophils

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Kuna, MD, Principal Investigator — University of Pennsylvania; Raymond R Townsend, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No